CLINICAL TRIAL: NCT00550810
Title: A Phase II Study of SU011248 for Maintenance Therapy in Hormone Refractory Prostate Cancer After First Line Chemotherapy
Brief Title: Sutent Maintenance After Response to Taxotere
Acronym: SMART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alberta Health services (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Rachel Syme, Dr. Bernie Eigl, Alberta Health services
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBCC-0707001; SMART
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-09

CONDITIONS: Prostate Cancer; Hormone Refractory
Keywords: Sutent
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sunitinib (SU011248) — SU011248 (study medication) will be given at 50 mg/day as a single agent for 4 consecutive weeks followed by a 2 week rest period to form a complete cycle of 6 weeks. Study medication will be orally self administered once daily without regard to meals beginning on Day 1 of the study. Cycles will be repeated in the absence of unacceptable toxicity or disease progression
  Other Names: Sutent

SUMMARY:
The major goal is to determine whether the experimental agent has clinically promising activity that would merit progression to a formal phase III trial.

Patients with hormone refractory prostate cancer after docetaxel chemotherapy have limited treatment options and no systemic treatment has been proven to be effective. Because of its action, safety and simple administration SU011248 has potential for effectiveness in this disease setting. Promising activity in this study would provide the necessary proof-of-principle for a larger confirmatory study in this population, and potentially in earlier stages of this common disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of adenocarcinoma of the prostate
* Metastatic or locally recurrent disease not curable with standard therapy
* ECOG performance status 0, 1 or 2
* Prior single agent docetaxel or docetaxel combination chemotherapy with a documented PSA or imaging response, and no objective evidence of disease progression at study enrolment

Exclusion Criteria:

* Patients with a history of other invasive cancer, except adequately treated non
* melanoma skin cancer.
* Patients with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SU011248.
* Other serious intercurrent illness or medical condition that might be aggravated by protocol treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 180 days without evidence of disease progression would be considered clinically worthy of further investigation

SECONDARY OUTCOMES:
-PSA Response -Toxicity | The secondary endpoint of PSA response will also be documented. PSA response is defined as a ≥50% fall in PSA (minimum of 5 µg/L) from baseline maintained for > 3 weeks and without evidence of disease progression otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Eigl, M.D., Study Chair — Tom Baker Cancer Board
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario